CLINICAL TRIAL: NCT00805896
Title: Effectiveness and Safety Study of TACE Plus Oral Songyou Granule for Unresectable HCC
Brief Title: Songyou Granule and Transarterial Chemoembolization for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Boheng Zhang/Liver Cancer Institute, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCI-1001
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Hepatocellular Carcinoma; Unresectable
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — songyou yin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Songyou Granule
  Interventions: Drug: Songyou
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Songyou — 4g/pack
  Arms: 1
Drug: placebo — 4g/pack
  Arms: 2

SUMMARY:
Songyou Granule is a mixture of 6 herbs. Vitro and vivo studies showed that Songyou Granule can inhibit HCC cells grow, and HCC metastasis. Hypothesis of this study is that TACE plus Songyou Granule will improve outcome in patients with advanced hepatocellular carcinoma (HCC) compared with TACE.

DETAILED DESCRIPTION:
Primary outcome Measures:

To evaluate the effect of TACE plus Songyou Granule or TACE plus placebo on TTP

Secondary Outcome Measures:

* Overall survival (OS)
* Progression Free Survival (PFS)
* The overall response rate
* Time to symptomatic Progression
* In an exploratory manner the relative TTP, TTSP, RR and overall survival between the 2 study populations
* Overall response duration and time to objective response
* Overall disease control rate
* The safety, tolerability, and adverse event profiles of the two treatment regimens used in this trial

Enrollment: 260 Study Start Date: January 2009 Study Completion Date: December 2010 Primary Completion Date: December 2010 (Final data collection date for primary outcome measure)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (≥ 18 years of age) with a diagnosis of HCC which is not amenable to surgical resection or local ablative therapy
* Histological confirmed HCC or clinical/laboratory diagnosis of HCC or nodules larger than 2 cm with typical vascular features or AFP > 200
* Patient must have quantifiable disease limited to the liver
* Patients must have at least one tumor lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to RECIST criteria
  * The lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* ECOG performance status (PS) <2
* No prior targeted antiangiogenic therapy. Metronomic chemotherapies are allowed. At least 4 weeks since prior systemic chemotherapy
* No significant baseline liver dysfunction. Cirrhotic status of Child-Pugh class A or B
* No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
* The following laboratory parameters:

  * Platelet count ≥ 50,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 2 mg/dL
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or a PTT within normal limits
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC except cervical carcinoma in situ, treated basal-cell carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), and any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring hemo- or peritoneal dialysis
* Child-Pugh C hepatic impairment
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Known central nervous system tumors including metastatic brain disease
* History of organ allograft
* Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Patients unable to swallow oral medications.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of the study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Time to tumor progression(TTP) | Dec 2008 to Dec 2010

SECONDARY OUTCOMES:
Overall survival (OS) | Dec 2008 to Dec 2010

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-You Tang, MD, Study Chair — Fudan University; Boheng Zhang, MD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Liver Cancer Institute and Zhongshan Hospital, Shanghai, Shanghai Municipality